CLINICAL TRIAL: NCT01139242
Title: Increasing CRC Screening in Urban African American Communities Via Churches
Brief Title: Increasing Colorectal Cancer Screening in Urban African American Communities Via Churches
Acronym: ACTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-1271; U48DP000059-02S1 (NIH)
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2010-06

CONDITIONS: Colorectal Cancer
Keywords: CRC screening status; physical activity level; fruit and vegetable consumption; Early Detection of Cancer; Colorectal Cancer (CRC) screening status
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Body & Soul nutritional intervention (Other): This is a standardized intervention to increase fruit and vegetable consumption among church members through pastoral and peer counseling and church activities/menus.
  Interventions: Behavioral: Body & Soul nutritional intervention
- Newsletters/peer counseling (Experimental): Four tailored newsletters and peer counseling calls to promote CRC screening among church members out-of-date according to screening guidelines. For those up-to-date, promotion is of increased physical activity.
  Interventions: Behavioral: Experimental: newsletters and peer counseling

INTERVENTIONS:
Behavioral: Body & Soul nutritional intervention — Pastoral and peer counseling, and church activities/menus to promote increased fruit and vegetable consumption among church members.
  Arms: Body & Soul nutritional intervention
Behavioral: Experimental: newsletters and peer counseling — Four tailored newsletters and peer counseling calls to promote CRC screening in church members who are out-of-date with screening. Four tailored newsletters and peer counseling calls to others to increase physical activity.
  Arms: Newsletters/peer counseling

SUMMARY:
This is an intervention study to increase colorectal cancer screening and physical activity in members of African-American churches who are 50 years old and older. The control arm receives the Body & Soul program, a program to increase fruit and vegetable intake. The investigators hypothesize that those receiving the intervention, which includes four tailored newsletters and peer counseling, will be more likely to be screened if not up-to-date, and more likely to increase physical activity if screening was up-to-date at baseline, than controls.

ELIGIBILITY:
Inclusion Criteria:

* Members of African-American churches who are at least 50 years old.

Exclusion Criteria:

* Non-members of African-American churches; members who are under 50 years of age.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 955 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Higher incidence of CRC screening, if needed, among experimental participants. | One year
  Among church members who were out-of-date for CRC screening at baseline, a higher percentage of experimental participants will have been screened at the time of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Marci K Campbell, PhD, Principal Investigator — UNC - Chapel Hill